CLINICAL TRIAL: NCT01610583
Title: Development of a Tool to Assess Spanish-Language Genetic Literacy
Brief Title: Testing Spanish-language Genetic Literacy
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912144; 12-HG-N144
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-02-23

CONDITIONS: Genetic Literacy
Keywords: Genetic Literacy; Latino

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Health literacy means being able to understand basic health care information. This information can include drug labels and prescription instructions. It can also include doctor s instructions. Better health literacy can help improve a person s health outcomes.
* Many minorities have low health literacy. Latinos in particular have both low health literacy and poor health outcomes. Language barriers such as poor reading skills can contribute to problems with health literacy. Researchers want to develop a new health literacy measuring tool. This tool will focus on genetic literacy, which involves understanding personal risk of health problems. The tool will be written in Spanish. The study will work with Spanish-speaking Latinos to develop and test this genetic literacy tool.

Objectives:

- To develop a Spanish-language tool to study genetic literacy.

Eligibility:

- Spanish-speaking Latino adults between 18 and 75 years of age.

Design:

* Participants will be screened with a brief interview. No personal samples will be needed.
* Participants will complete the genetic literacy questionnaire. It will be given in Spanish.
* The tool will ask about participants personal and family health history. It will also ask about their understanding of genetic terms and genetic testing. Other personal information, such as level of education, will be collected.
* Participants will receive a gift card for completing the survey.
* No treatment or genetic counseling will be provided as part of this study.

DETAILED DESCRIPTION:
The proposed study seeks to better understand genetic literacy in the U.S. Latino

population by developing and validating a Spanish-language measure of genetic literacy and

subsequently exploring the relationships between genetic literacy, personal characteristics,

exposure to genetics, acculturation, and self-efficacy to discuss family health history

information. This study is primarily informed by research in health literacy, which is defined as

an individual s ability to understand and use health information to make informed decisions.

Past research has modeled the effects of demographic factors, prior experience, and prior

knowledge on health literacy, and in turn to health behaviors and outcomes. These same

domains apply when considering the concept and operationalization of genetic literacy: an

individual s ability to understand and use genetics-related information to make informed

decisions.

Numerous studies have reported the wide prevalence of disparities among minorities in various areas of healthcare, including use of genetics services, and many of these inequalities have been related to low health literacy. Latinos represent one group in particular that has been shown to have both low health literacy and some of the poorest health outcomes. A few studies have explored the public s knowledge of genetics, and differences in level of understanding were found amongst minority groups. Given the increasing importance of genetics in healthcare and the rapidly growing population of Latinos in the U.S., it is of particular importance to assess this population s genetic literacy. The first aim of this study is to develop a Spanish-language genetic literacy measure and validate it against an existing Spanish-language health literacy measure. Then this study will examine the relationship of genetic literacy in the Latino population to certain demographic characteristics, previous exposure to genetics, acculturation, and participants self-efficacy to discuss health history information with family members and providers. Study participants will be recruited through convenience sampling in three different areas of Maryland with a high percentage of Latinos. This study will contribute to the limited body of knowledge about genetic literacy in the Latino population, and expand understanding of how genetic literacy influences individuals genetics-related self-efficacy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants eligible for this study will include all Spanish-speaking Latino males and females between 18 and 75 years of age (self-reported) recruited in the Baltimore, MD,

Montgomery County, MD, or Prince George s County, MD areas. Individuals do not have to be Maryland residents, as recruitment for this study will be conducted through convenience sampling.

-Participants must self-report Spanish as their primary language and therefore have limited English fluency.

EXCLUSION CRITERIA:

* Individuals over the age of 75 will be excluded because there is a possibility of confounding between literacy and cognitive decline.
* Individuals under the age of 18 will be excluded because they are likely to have different genetic literacy levels than their adult counterparts due to different levels of exposure to genetics in school curriculums.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-05-24; Study Completion 2015-02-23

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baker DW. The meaning and the measure of health literacy. J Gen Intern Med. 2006 Aug;21(8):878-83. doi: 10.1111/j.1525-1497.2006.00540.x. No abstract available. PMID 16881951
- [Background] Bowling BV, Acra EE, Wang L, Myers MF, Dean GE, Markle GC, Moskalik CL, Huether CA. Development and evaluation of a genetics literacy assessment instrument for undergraduates. Genetics. 2008 Jan;178(1):15-22. doi: 10.1534/genetics.107.079533. PMID 18202354
- [Background] Davis TC, Crouch MA, Long SW, Jackson RH, Bates P, George RB, Bairnsfather LE. Rapid assessment of literacy levels of adult primary care patients. Fam Med. 1991 Aug;23(6):433-5. PMID 1936717